CLINICAL TRIAL: NCT05010889
Title: Health-Related Quality of Life After Peroral Endoscopic Myotomy for Patients With Achalasia
Brief Title: Quality of Life After POEM for Achalasia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Xiangbin Xing, Principal Investigator, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: 124
Record Dates: First submitted 2021-08-10; First posted 2021-08-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Esophageal Achalasia
Keywords: Esophageal Achalasia, Peroral Endoscopic Myotomy, Quality of Life
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Achalasia patients: Patients schedule to undergo POEM for treatment of symptomatic achalasia. The diagnosis of achalasia was based on high resolution manometry, barium esophagram, and upper endoscopy.
  Interventions: Procedure: Peroral endoscopic myotomy (POEM)

INTERVENTIONS:
Procedure: Peroral endoscopic myotomy (POEM) — POEM is performed as previously described by Inoue et al (Endoscopy 2010), including four main steps mucosal incision, submucosal tunneling, myotomy and mucosal entry closure.

SUMMARY:
Achalasia is an esophageal motility disorder, characterized by insufficient lower esophageal sphincter relaxation and loss of esophageal peristalsis. Patients with achalasia experience distressing gastrointestinal symptoms, including dysphagia, reflux and chest pain, which lead to weight loss and malnutrition. Undoubtedly, health-related quality of life can be significantly diminished in patients with achalasia. At present, POEM has become one of the standard therapies for achalasia. Limited studies have focused on the patient's quality of life before and after POEM. The present study aimed to assess the changes in quality of life of patients with achalasia using the validated achalasia severity questionnaire (ASQ) and the short form (SF)-36 scale.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as achalasia base on high resolution manometry, barium esophagram and upper endoscopy
* Scheduled to undergo POEM for treatment of achalasia

Exclusion Criteria:

* Coagulopathy and systemic disorders that precluded safe general anesthesia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients schedule to undergo POEM for treatment of symptomatic achalasia in one tertiary hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Achalasia symptom questionnaire (ASQ) | Baseline, Change from Baseline ASQ score at 3 months and 12 months after treatment
  Achalasia symptom questionnaire assess the disease-specific health-related quality of life by sampling the concepts of food tolerance, dysphagia-related behavior modifications, pain, heartburn, distress, lifestyle limitation, and satisfaction in 10 items. The total range is 10 to 31, with higher scores indicating worse quality of life (Urbach et al, Am J Gastroenterol 2005).
Short form (SF)-36 | Baseline, Change from Baseline SF-36 score at 3 months and 12 months after treatment
  The short form (SF)-36 (best score 100, worst score 0). The short form (SF)-36 assess the health-related quality of life from 8 aspects, including physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional and mental health in 36 items. The total range is 0 to 100, with lower scores indicating worse quality of life (Ware et al, J Clin Epidemiol 1998).

SECONDARY OUTCOMES:
Eckardt score | baseline, 3 months and 12 months after treatment
  The Eckardt score assesses the severity of achalasia symptoms by combining the sum of symptom frequency scores for dysphagia, regurgitation, and chest pain and a weight loss score. Each component can be graded from 0 to 3 points. The total range is 0 to 12, with higher scores indicating more severe symptoms (Eckardt AJ et al, Nat Rev Gastroenterol Hepatol 2011).
Gastroesophageal reflux disease questionnaire (GerdQ) score | baseline, 3 months and 12 months after treatment
  The GerdQ has been developed as a tool to facilitate the symptom-based diagnosis of GERD. Scores ranging from 0 to 3 were applied for the four positive predictors (heartburn, regurgitation, sleep disturbance due to reflux symptoms and use of over-the-counter medications for reflux symptoms) and from 3 to 0 for two negative predictors (epigastric pain and nausea). The GerdQ score was calculated as the sum of these scores, giving a total score ranging from 0 to 18. A total GerdQ score >7 is considered indicative of significant GERD symptoms (Jones R et al, Aliment Pharmacol Ther 2009).
Reflux esophagitis on post-POEM endoscopy | 3 months after treatment
  The severity of reflux esophagitis is graded according to the Los Angeles classification (Armstrong D et al, Gastroenterology 1996).

CONTACTS AND LOCATIONS:
Overall Officials: Xiangbin Xing, MD, PhD, Study Director — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No